CLINICAL TRIAL: NCT03278535
Title: Reference Gait Data for Healthy Subjects: Caren-based Gait Analysis
Brief Title: Reference Gait Data for Healthy Subjects
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL61229.068.17
Record Dates: First submitted 2017-07-11; First posted 2017-09-11 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-07

CONDITIONS: Healthy Subjects; Healthy Volunteers; Healthy Adults

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- age group 18-29 years: CAREN-based gait analysis: 20 men and 20 women aged between 18-29 years
  Interventions: Diagnostic Test: CAREN-based gait analysis
- age group 30-39years: CAREN-based gait analysis: 20 men and 20 women aged between 30-39years
  Interventions: Diagnostic Test: CAREN-based gait analysis
- age group 40-49years: CAREN-based gait analysis: 20 men and 20 women aged between 40-49years
  Interventions: Diagnostic Test: CAREN-based gait analysis
- age group 50-59years: CAREN-based gait analysis: 20 men and 20 women aged between 50-59years
  Interventions: Diagnostic Test: CAREN-based gait analysis
- age group 60-69years: CAREN-based gait analysis: 20 men and 20 women aged between 60-69years
  Interventions: Diagnostic Test: CAREN-based gait analysis
- age group 70+: CAREN-based gait analysis: 20 men and 20 women aged between 70 years and older
  Interventions: Diagnostic Test: CAREN-based gait analysis

INTERVENTIONS:
Diagnostic Test: CAREN-based gait analysis — subjects only walk at CAREN at different speed

SUMMARY:
Three dimensional gait analysis is widely accepted as a general measure of functional ability among individuals as it is related to health, well-being and quality of life. To diagnose subtle changes/deviations in gait and to correctly interpret gait, a reference gait database of healthy subjects is required. Computer Assisted Rehabilitation Environment (Caren) is a new gait analysis system which combines the 3D motion captures system with a split belt force plate instrumented treadmill and a virtual reality environment. This system enables to analyses several successive steps, which is impossible in the standard overground laboratories. Until now, no reference gait database has been created using the Caren system. The aim of this descriptive study is to create a reference database of gait in healthy adults with varying subject characteristics using Caren. This study is a single center descriptive study to build a reference database on gait of healthy adults of different ages. Six age groups are composed existing of 20 males and 20 females. Taken into account that 10% of the volunteers (especially elderly) may drop out due to e.g. disability, a total of 264 subjects will be recruited to ensure that database will include 240 subjects. Inclusion criteria: ambulatory, ability to walk without aid for 30 minutes, age older than 18 years and willing to participate. Exclusion criteria: muscular skeletal, cardiopulmonary disorders or other diseases significantly influencing gait. Medical interventions, such as surgical treatment or botulinium toxin 6 months, which significantly influence gait. Subjects will walk at different walking speeds at Caren while gait is measured. Subjects always wear a safety harness to avoid falling. In addition adults wear standard shoes (gymnastic booties) provided by the lab to avoid shoes effects. All subjects undergo measurement of leg length, body length and body weight in order to retrieve anthropometric parameters. In addition a standard physical examination is performed to get information about a subjects' muscle strength, balance and articular mobility of the hip, knee and ankle. Gait kinematic, kinetic, spatio-temporal and balance parameters are measured.

DETAILED DESCRIPTION:
Gait is one of the most important activity of daily life for humans. In clinical and research settings, gait performance is widely accepted as a general measure of functional ability among individuals. Computer Assisted Rehabilitation ENvironment (CAREN; Motek Medical, Amsterdam, The Netherlands) is a relatively novel system to analyze gait in a safe and accurate way. CAREN consists of an instrumented split-belt treadmill mounted onto a 6-degree-of-freedom motion platform in combination with a Virtual Environment projected on a 180° semi-cylindrical screen. Two force plates underneath each belt and 12 3D motion capture cameras (VICON system) allow an accurate analysis of gait which is expressed by kinematic, kinetic, spatiotemporal en dynamic balance parameters. Currently at the MUMC+, CAREN-based gait analysis is used for clinical purposes and is increasingly more applied to contribute in clinical diagnostics and decision-making and to evaluate interventions and rehabilitation programs. Besides, the CAREN system is applied in gait analysis laboratory settings as an alternative or an additive to over ground gait analysis. However, due to its novelty, size, high costs, and complexity, the CAREN system is not a widely accessible technology. Literature is limited and research is still in progress. From these experiences, it is known that CAREN is safe in use.

An individuals' walking pattern is variable and can change due to several factors such as advancing age. Furthermore gait is influenced by body characteristics such sex, body height and mass. Gait also changes as a result of health-related factors such as pain and diseases. Moreover gait can change through rehabilitation and training. This all suggests that human gait analysis is useful for clinical purposes, for example for diagnostics or to evaluate rehabilitation programs. However to apply human gait analysis in clinical practice, it is crucial to have insight into the normal walking pattern of individuals. A gait database of healthy subjects with varying subject characteristics (e.g. age) is required to ensures that gait is correctly interpreted. This database will give further insight in the dynamics of walking, clarifying the level and proportion in which gait is affected by subject characteristics and walking speed. This insight will improve the interpretation of gait, and thus contribute to improved clinical diagnostics and follow up capabilities. In addition the database will be relevant in clinical practice as it quickly puts into perspective gait of patients. Moreover it enables the detection of subtle changes in gait (e.g. after intervention).

Objective and hypothesis:

This research is a single center descriptive study to create a reference database of gait of healthy adults of different ages. Six age groups are composed (18-29yrs, 30-39yrs, 40-49yrs, 50-59yrs, 60-69yrs, >70yrs), existing of 20 males and 20 females.

This descriptive study aims to build a reference gait database for healthy subjects based on CAREN including kinematic, kinetic, spatio-temporal and balance parameters. Values for gait parameters of healthy adults will be created for varying age groups and sex. In addition, knowing the impact of walking speed on various gait parameters, gait parameters of healthy subjects will be clustered per walking speed, taking sex and age into account.

Primary Objective:

A descriptive study to collect a Caren-based reference database for healthy gait.

Secondary Objectives:

* To investigate effects of subject characteristics such as age, sex and leg length on gait kinematic, kinetic, temporal-spatial and balance parameters.
* To investigate the relation between walking speed and gait kinematic, kinetic, temporal-spatial and balance parameters.

Methods:

This is a single center descriptive study performed at the department Physiotherapy of the Maastricht University Medical Center (MUMC+) in which gait of healthy adult volunteers of varying ages is obtained by the new Computer Assisted Rehabilitation ENvironment (Caren) system. The collected data will be used to create a database for gait parameters of healthy subjects.

120 healthy men and 120 healthy women, equally divided over the six age groups (18-29j, 30-39j, 40-49j, 50-59j, 60-69j, >70j) are included.

The healthy adult volunteers will walk at different walking speeds at the Caren system.

First, the comfortable walking speed of the subject is determined using a ramp protocol. This includes that subject starts walking at 0.5m/s and that the speed is increased every second by 0.01m/s until the subject reached the comfortable walking speed. This is repeated 3 times. The average of these 3 walking speeds is used as comfortable walking speed. Afterward, the subject walks for 5 minutes at the fixed comfortable speed to get familiarized to the system. After familiarization, the measurement starts. The volunteers will walk at comfortable speed, at a slow speed (comfortable speed - 30%), a fast speed (comfortable speed + 30%) and at a slower speed (fixed at 0.5km/h). These four conditions are randomly applied to eliminate a possible effect of sequence of performed walking speed (and thus familiarization) on gait. Every measurement is proceeded by a 2 minute habituation period at that specific walking speed. Subjects will wear a safety harness to avoid falling. In addition adults wear standard shoes (gymnastic booties) provided by the lab to avoid shoes effects.

Gait kinematics (joint angles), kinetics (joint moments and power), spatio-temporal parameters (e.g. stride length) and dynamic balance parameters (e.g. margins of stability) will be determined. Values for gait parameters of healthy adults will be created and clustered for varying age groups, sex and walking speeds.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory
* Ability to walk without aid for 30 minute
* Willing to participate and able to provide informed consent.
* 18 years or older

Exclusion Criteria:

* Muscular skeletal, cardiopulmonary disorders or other diseases significantly influencing gait.
* Medical interventions, such as surgical treatment or botulinium toxin 6 months, which significantly influence gait.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The aim of the study is to create a reference database consisting of 240 healthy (120 men, 120 women), ranging from 18 years to > 70yrs. For each of the six age categories (18-29yrs, 30-39yrs, 40-49yrs, 50-59yrs, 60-69yrs, >70yrs), 20 men and 20 women will be included. Assuming that 10% of the volunteers (especially elderly) may drop out because subjects cannot complete the protocol due to fatigue, impaired condition, fear etc., an additional 10% will be recruited to ensure that 240 subjects will be included at the end. This results in a total of 264 subjects that will be recruited. When subjects do not want to continue participating in the study and want to stop the procedure, the subjects can stop at any time and withdraw without any reason.
Sampling Method: Non-Probability Sample
Enrollment: 264 (Actual)
Dates: Start 2017-07-04 (Actual); Primary Completion 2021-06-03 (Actual); Study Completion 2021-06-03 (Actual)

PRIMARY OUTCOMES:
CAREN-based kinematic gait parameters | 4-7-2017 until 3-6-2021
  Kinematics of the hip, knee and ankle measured during the gait cycle (e.g. stance phase knee flexion).
CAREN-based kinetic gait parameters | 4-7-2017 until 3-6-2021
  Kinetics of the hip, knee and ankle measured during the gait cycle (e.g. flexion/extension moments of the hip)
CAREN-based spatiotemporal gait parameters | 4-7-2017 until 3-6-2021
  e.g. walking speed, stride time, cadence, step width, step length.
CAREN-based balance parameter | 4-7-2017 until 3-6-2021
  mediolateral and backward margins of stability (MoS)

SECONDARY OUTCOMES:
anthropometric characteristic: body height | 4-7-2017 until 3-6-2021
  Body height (cm)
anthropometric characteristic: body weight | 4-7-2017 until 3-6-2021
  Body weight (kg)
anthropometric characteristic: leg length | 4-7-2017 until 3-6-2021
  Leg length (cm)

CONTACTS AND LOCATIONS:
Overall Officials: Rik Marcellis, Dr, Principal Investigator — Maastricht UMC - dept. Fysiotherapy
Locations (1):
- Maastricht UMC, Maastricht, Limburg, Netherlands